CLINICAL TRIAL: NCT01498263
Title: Inherited Diseases, Caregiving, and Social Networks
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120022; 12-HG-0022
Record Dates: First submitted 2011-12-21; First posted 2011-12-23 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-10-28

CONDITIONS: Undiagnosed Disease; Healthy Volunteer (Adult With Typically Developing Child); Inherited Neurodegenerative Disorders; Inherited Metabolic Disorders (Inborn Errors of Metabolism); Alzheimer's Disease and Related Dementias
Keywords: Genetic Condition; Family Network; Social Support; Natural History
MeSH Terms: conditions — Undiagnosed Diseases; Metabolism, Inborn Errors; Alzheimer Disease; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Alzheimers related dementias (family): Enrollment was open to family members of persons diagnosed with Alzheimers (/related dementia) in specific communities around Memphis, TN.
- Inherited inflammatory condition (family): Enrollment open to family members of persons diagnosed with inherited inflammatory conditions. Participation at NIH or remote (internet/phone); request referral of family for remote participation.
- Inherited metabolic conditions (family): Enrolls family members of persons diagnosed with inborn errors of metabolism / mitochondrial disorders. Study at NIH or remote (internet/phone); request family-referrals for remote participation.
- Inherited neurodegenerative disorders (family): Open to family members of persons diagnosed with genetically-defined neurodegenerative conditions. Study at NIH or (internet/phone); request referral of family members for remote participation.
- Typically developing (family) = Healthy Volunteers: Open to parents of typically-developing child/ren <18yrs (*when age-matched child is full-time resident of parent's home). Study at NIH; request family-referrals for remote participation.
- Undiagnosed conditions (family): Enrollment open to family members referred in from the Undiagnosed Disease Network. Participation at NIH or remote (internet/phone); request referral of family members for remote participation

SUMMARY:
Approximately 66 million informal caregivers care for someone who is ill, disabled, or aged. These caregivers experience significant distress associated with caregiving, which may be particularly salient in the context of inherited conditions. Previous studies have not examined caregiving from a network perspective, nor have they considered how cognitive and emotional responses, such as caregivers worry for themselves and relatives acquiring the disease or guilt related to the genetic etiology of their child s illness, as possible stressors; the current project fills this literature gap.

Caregiving processes may vary across type of illness and the life course. In illnesses that impact children, parents and grandparents may take on caregiving roles whereas in conditions that impact adults, spouses and adult children may provide care. Caregivers must adapt to the strain of caring for their affected relatives and this adaptation may differ depending on caregiver roles. The caregiver s support network may influence adaptation, impacting the health and well-being of patients, their caregivers, and other relatives.

This project, comprised of 5 substudies, will examine social contexts surrounding families involved in caring for individuals with chronic inherited conditions from a relational perspective. Surveys and interviews will assess participants cognitions and emotions about the disease, caregiving burden and caregiving/support network systems. In addition, biomarkers will be considered in 2 substudies to examine how caregiving roles and expectations impact health among caregivers. As part of our current inquiry, we have

developed an assessment tool aimed at understanding caregiver experiences related to dietary practices in the context of metabolic conditions. To evaluate the psychometric properties of this scale, we propose a fifth substudy under the current protocol.

We aim to recruit at least 5550 participants through residential/daycare centers, advocacy groups, and the NIH Clinical Center. We will recruit formal caregivers, multiple biological and non-biological adult relatives of affected individuals and typically developing controls to construct and evaluate caregiving/support network systems. This project will use a social network framework to develop and adapt common measures of caregiving roles to evaluate burden, perceptual bias, and unmet expectations in caregiving. The psychometric properties of these new measures, characteristics of family caregiving and support networks, and how these network characteristics are associated with caregiving strain and well-being, including biomarkers of physical health, will be investigated. The moderating role of family members cognitions and emotions and disease context will be considered. Findings will guide future research to develop network-based interventions promoting positive adaptation to the presence of inherited conditions in families through improved social environments and coping skills....

DETAILED DESCRIPTION:
Approximately 66 million informal caregivers care for someone who is ill, disabled, or aged. These caregivers experience significant distress associated with caregiving, which may be particularly salient in the context of inherited conditions. Previous studies have not examined caregiving from a network perspective, nor have they considered how cognitive and emotional responses, such as caregivers worry for themselves and relatives acquiring the disease or guilt related to the genetic etiology of their child s illness, as possible stressors; the current project fills this literature gap.

Caregiving processes may vary across type of illness and the life course. In illnesses that impact children, parents and grandparents may take on caregiving roles whereas in conditions that impact adults, spouses and adult children may provide care. Caregivers must adapt to the strain of caring for their affected relatives and this adaptation may differ depending on caregiver roles. The caregiver s support network may influence adaptation, impacting the health and well-being of patients, their caregivers, and other relatives.

This project, comprised of 5 substudies, will examine social contexts surrounding families involved in caring for individuals with chronic inherited conditions from a relational perspective. Surveys and interviews will assess participants cognitions and emotions about the disease, caregiving burden and caregiving/support network systems. In addition, biomarkers will be considered in 2 substudies to examine how caregiving roles and expectations impact health among caregivers. As part of our current inquiry, we have developed an assessment tool aimed at understanding caregiver experiences related to dietary practices in the context of metabolic conditions. To evaluate the psychometric properties of this scale, we propose a fifth substudy under the current protocol.

We aim to recruit at least 5550 participants through residential/daycare centers, advocacy groups, and the NIH Clinical Center. We will recruit formal caregivers, multiple biological and non-biological adult relatives of affected individuals and typically developing controls to construct and evaluate caregiving/support network systems. This project will use a social network framework to develop and adapt common measures of caregiving roles to evaluate burden, perceptual bias, and unmet expectations in caregiving. The psychometric properties of these new measures, characteristics of family caregiving and support networks, and how these network characteristics are associated with caregiving strain and well-being, including biomarkers of physical health, will be investigated. The moderating role of family members cognitions and emotions and disease context will be considered. Findings will guide future research to develop network-based interventions promoting positive adaptation to the presence of inherited conditions in families through improved social environments and coping skills.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Adult family members of the individuals affected by an inherited disease (e.g. Alzheimer s disease, inborn errors of metabolism and mitochondrial disease, lysosomal storage disorder, genetic neurodegenerative disorder, undiagnosed diseases, and inherited

inflammatory conditions) OR

* Informal caregivers of the affected individual OR
* Caregivers family members OR
* Formal caregivers who are identified as part of patients caregiving networks will be eligible for recruitment in the study OR
* For the control group in Substudy 2, adult family members of normally developing children, informal caregivers, caregivers family members and formal caregivers who are identified as part of the child s caregiving network will be eligible for recruitment in the study.

(For better matching across groups: in the Healthy Volunteer controls, the normally developing focus child must live in the parent/caregiver household on a full-time basis.)

* Participants are eligible for biospecimen collection in Substudies 3 only if two parents/caregivers are present in the household, eligible, and willing to provide biospecimens.
* Fluency in English

EXCLUSION CRITERIA:

* Those who are unable to complete the survey and interviews
* Affected individuals/Patients with condition being studied
* Individuals under the age of 18
* Those who have fever or signs of acute infection on the collection day, have been hospitalized in the past 3 months, and women who are currently pregnant or nursing will not be eligible for the biospecimen collection portion of Substudies 2 and 3 but will be eligible for the survey/interview portion of the substudies.
* Control group individuals will be excluded if they serve as a caregiver for anyone in their family affected by any major medical condition.
* Staff of NHGRI (National Human Genome Research Institute)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a study has family-based enrollment of caregivers and their social support networks. Specific context of recruitment may vary depending upon the health condition of the affected family member; number of severe, chronic conditions with genetic basis are among the inclusion criteria. For the substudy of caregivers of persons affected by Alzheimer s disease and related dementias (AD), recruitment took place in residential facilities in Memphis, TN [substudy1; data analysis only]. Caregivers of persons affected by inborn errors of metabolism, genetic neurodegenerative conditions, or with severe chronic undiagnosed conditions may be referred in to the protocol by NIH collaborators or through advocacy groups. Healthy volunteers (parents of healthy child/ren) are recruited through NIH and in the community. The study uses snowball sampling of self-referral: each participant is invited to refer in support network members who also provide support/care for the focus-relative.
Sampling Method: Non-Probability Sample
Enrollment: 682 (Actual)
Dates: Start 2012-01-09 (Actual)

PRIMARY OUTCOMES:
Measures of caregiving processes | Interim, completion
  Develop measures of caregiving processes within family social network systems
Family network characteristics | Interim, completion
  Identify family network characteristics associated with positive adaptation

CONTACTS AND LOCATIONS:
Overall Officials: Laura M Koehly, Ph.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - University of Memphis, Memphis, Tennessee

REFERENCES:
- [Derived] Zajdel M, Davidson H, Lea D, Koehly LM. Links of we-talk to caregiver social network systems and health. J Fam Psychol. 2022 Dec;36(8):1386-1396. doi: 10.1037/fam0001013. Epub 2022 Aug 4. PMID 35925717
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-HG-0022.html